CLINICAL TRIAL: NCT05745376
Title: Addressing Disparities in Food Access Among Young Children in Louisiana: A Farm to ECE Approach
Acronym: FarmtoECE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xavier University of Louisiana. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB881-23
Record Dates: First submitted 2023-02-06; First posted 2023-02-27 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Food Insecurity; Health Knowledge, Attitudes, Practice; Nutrition, Healthy
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Intervention Model Description: intervention and comparison
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Center (Experimental): The intervention will include: (1) assisting ECEs with conducting self-assessments; (2) connecting ECEs with local farmers and food producers; (3) providing technical assistance for menu changes, procuring healthy food, identifying and implementing best feeding practices and policies for the environment; (4) delivering nutrition education; and (5) connecting parents/guardians with local food resources and affordable fresh food to be consumed at home
  Interventions: Behavioral: Farm to ECE programming
- Comparison (No Intervention): No programming at center, only surveys

INTERVENTIONS:
Behavioral: Farm to ECE programming — Students and parents at this center will receive program elements described in arm descriptions.
  Arms: Intervention Center

SUMMARY:
The goal of this pilot project is to increase access to healthy food, improve diets, and reduce food insecurity and, in turn, reduce health disparities among low-income, minority children under the age of five attending early childcare centers. Specific aims are to: 1) examine the feasibility of a six-month Farm to ECE intervention and 2) collect preliminary data to evaluate the efficacy of the program to 2.1) improve the ECE nutrition environment from baseline to follow-up; 2.2) increase access to local fruits and vegetables among children at ECEs from baseline to follow-up; and 2.3) increase parent knowledge and use of community food resources. The investigators will use this preliminary data to develop a larger scale project to test intervention efficacy.

DETAILED DESCRIPTION:
The pilot study will take place at four centers within a network of Catholic Charities Early Head Start and Head Start Centers in New Orleans, Louisiana. Two centers will serve as intervention sites and two as comparison sites. Over 90% of the network centers' students identify as Black, and all qualify for federally funded free meals and snacks. The intervention will include: (1) assisting ECEs with conducting self-assessments; (2) connecting ECEs with local farmers and food producers; (3) providing technical assistance for menu changes, procuring healthy food, identifying and implementing best feeding practices and policies for the environment; (4) delivering nutrition education; and (5) connecting parents/guardians with local food resources and affordable fresh food to be consumed at home. The intervention will be implemented for 6 months.

Aim 1 uses a cross-sectional mixed methods design, collecting both quantitative and qualitative data in intervention centers. Aim 2 uses a pre-post design with a comparison group, collecting quantitative survey data at the center and parent level. At baseline and six-month follow-up, the investigators will conduct short surveys with staff and parents/caregivers of children attending ECEs.

ELIGIBILITY:
Inclusion Criteria (Key informant interviews and center assessments):

* Director or staff of participating center
* 18 years of age minimum

Exclusion Criteria (Key informant interviews and center assessments):

• Staff not involved with educational programming

Inclusion Criteria (Parent/guardian surveys):

* Parent or guardian of current student at participating center
* 18 years of age minimum

Exclusion Criteria (Parent/guardian surveys):

• None

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
incidence of parent/guardian use of community food resources | 6 months
  Parent/guardian surveys will ask questions about use of community food resources. Frequencies will be calculated based on results.
nutrition environment score measured by NAPSACC | 6 months
  Environmental assessments and pre/post staff surveys using validated tools (Nutrition and Physical Activity Self-Assessment for Child Care NAPSACC) will be used to determine changes in the nutrition environment and healthy options. Nutrition environment scores will be calculated using the tool scoring guide.
percent completion of program components (fidelity) | 6 months
  Staff will be asked to complete tracking records of all executed program components. Percent completion will be calculated by dividing program components executed by total program components.
satisfaction score with program implementation | 6 months
  Staff will be asked to complete a post intervention survey to indicate their satisfaction (scale of 1-5) with the program implementation and its components.

CONTACTS AND LOCATIONS:
Overall Officials: Megan Knapp, PhD, Principal Investigator — Xavier University of Louisiana.
Locations (1):
- Xavier University Of Louisiana, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No